CLINICAL TRIAL: NCT00831454
Title: Relationship of Polymorphisms and Mutations of Epidermal Growth Factor Receptor and Tyrosine Kinase Inhibitors Responsiveness in Non-small-cell Lung Cancer Patients
Brief Title: Identification of EGFR-TKIs Sensitivity or Resistance Markers in NSCLC May Help in Optimal Patient Selection
Status: Completed | Type: Observational
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Other Study IDs: ONC/OSS-02/2008
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: NON-SMALL-CELL LUNG CANCER
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to retrospectively evaluate associations between EGFR and AKT DNA-polymorphisms involved in transcriptional regulation and overall survival in NSCLC patients treated with EGFR-TKIs.

DETAILED DESCRIPTION:
DNA will be isolated from blood samples or paraffin-embedded tumor specimens and than a mutation analysis and SNPs genotyping will be done.

ELIGIBILITY:
Inclusion Criteria:

* Availability of tumor tissue or blood samples.
* Diagnosis of NSCLC
* At least one treatment with EGFR-TKIs inhibitors

Exclusion Criteria:

* Other than NSCLC primary diagnosis
* No treatment with EGFR-TKIs inhibitors
* No archival tissue available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NON-SMALL-CELL LUNG CANCER patients treated with EGFR-TKIs
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
to evaluate the presence of EGFR- and AKT-DNA polymorphisms. | At the end of enrollment

SECONDARY OUTCOMES:
to correlate the biological characteristics with clinical characteristics and survival data of patients. | At the end of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinco Humanitas, Rozzano, Mialno, Italy